CLINICAL TRIAL: NCT01330433
Title: Effects of CoSeal in Reducing Perioperative Bleeding & Adhesions in Pediatric Heart Surgery
Brief Title: Effects of CoSeal on Bleeding & Adhesions in Pediatric Heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Nahidh Hasaniya, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5110074
Record Dates: First submitted 2011-03-31; First posted 2011-04-07 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Congenital Heart Defect; Surgery-Induced Tissue Adhesions; Hemorrhage
MeSH Terms: conditions — Heart Defects, Congenital; Tissue Adhesions; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No CoSeal Surgical Spray (No Intervention): A patient randomized to the No CoSeal Surgical Spray group will not have CoSeal Surgical Spray applied at the end of their first staged procedure.
- CoSeal Spray Group (Experimental): CoSeal Spray will be applied at the end of the first staged procedure in patients randomized to the experimental group.
  Interventions: Device: CoSeal Surgical Spray Group

INTERVENTIONS:
Device: CoSeal Surgical Spray Group — A patient randomized to the CoSeal treatment group will have CoSeal Surgical Spray applied at the end of their first staged procedure.
  The dose regimen is as follows:
  * Patients weighing < 3kg will receive 1ml of CoSeal
  * Patients weighing 3-10kg will receive 1-2ml of CoSeal
  * Patients weighing >10kg will receive 2-4ml of CoSeal
  Arms: CoSeal Spray Group

SUMMARY:
This is a prospective, randomized, open-label, blinded-evaluator study that will evaluate the effectiveness of a surgical sealant (CoSeal) composed of biocompatible polyethylene glycol on the formation of mediastinal and pericardial adhesions in children undergoing staged surgical reconstruction (potential procedures include: Blalock-Taussig Type Operation, Classical Glenn Procedure, Bidirectional Glenn Procedure, Norwood). Additionally, bleeding will be evaluated by drainage post-operatively through surgical site drainage output.

ELIGIBILITY:
Inclusion Criteria:

* Have an acceptable surrogate capable of giving consent on the subject's behalf.
* Pediatric patients ages 0 - 17
* Have a cardiac disease which requires staged cardiac surgery and resternotomy
* Non-emergent state or emergent state with sufficient time to educate and consent

Exclusion Criteria:

* An immune system disorder
* Unplanned reoperation
* Known hypersensitivity to components in CoSeal
* Patients undergoing reoperation less than 3 months after the primary surgery

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nahidh Hasaniya, MD, Principal Investigator — Loma Linda University Medical Center; Anees Razzouk, MD, Study Chair — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CoSeal Spray Group: CoSeal Spray will be applied at the end of the first staged procedure in patients randomized to the experimental group.
  CoSeal Surgical Spray Group: A patient randomized to the CoSeal treatment group will have CoSeal Surgical Spray applied at the end of their first staged procedure.
  The dose regimen is as follows:
  * Patients weighing < 3kg will receive 1ml of CoSeal
  * Patients weighing 3-10kg will receive 1-2ml of CoSeal
  * Patients weighing >10kg will receive 2-4ml of CoSeal
Period: Overall Study
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Started | 16 | 19
Completed | 14 | 16
Not Completed | 2 | 3
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 19 | 35
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
Gender [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Severity of Adhesions at the Retrosternal Site
Description: Severity of adhesions at seven predefined sites (pericardial or retrosternal, inferior or diaphragmatic region, right lateral or arterial region, region around great vessels). Severity of adhesions is graded as 0 = no adhesions, 1 = filmy and avascular, 2 = requiring blunt dissection, 3 = requiring sharp dissection, 4 = requiring extensive sharp dissection. Adhesion scores for each patient will be derived from the sum of adhesion severity scores at each site, from 0 (no adhesions) to 28 (cohesive adhesions at all sites).
Time Frame: Severity of adhesions data will be collected during approximately the first 30-60 minutes of the second staged surgery
Measure: Number; unit: percentage of participants
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
percentage of participants
  no adhesions | 0 | 31.3
  filmy and avascular | 0 | 37.5
  requiring blunt dissection | 0 | 18.8
  requiring sharp dissection | 78.6 | 6.3
  requiring extensive sharp dissection | 21.4 | 6.3

2. Primary Outcome: Severity of Adhesions at the Arterial Base Site.
Description: Severity of adhesions at five predefined sites (retrosternal, diaphragmatic region, right lateral, left lateral, arterial base). Severity of adhesions is graded as 0 = no adhesions, 1 = filmy and avascular, 2 = requiring blunt dissection, 3 = requiring sharp dissection, 4 = requiring extensive sharp dissection. Adhesion scores for each patient will be derived from the sum of adhesion severity scores at each site, from 0 (no adhesions) to 28 (cohesive adhesions at all sites).
Time Frame: Severity of adhesions data will be collected during approximately the first 30-60 minutes of the second staged surgery
Measure: Number; unit: percentage of participants
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
percentage of participants
  no adhesions | 0 | 12.5
  filmy and avascular | 0 | 43.8
  requiring blunt dissection | 7.1 | 25.0
  requiring sharp dissection | 57.1 | 18.8
  requiring extensive sharp dissection | 35.7 | 0.0

3. Primary Outcome: Severity of Adhesions at the Diaphragm Site
Description: as for outcome 2
Time Frame: Severity of adhesions data will be collected during approximately the first 30-60 minutes of the second staged surgery
Measure: Number; unit: percentage of participants
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
percentage of participants
  no adhesions | 0 | 0
  filmy and avascular | 0 | 85.7
  requiring blunt dissection | 0 | 14.3
  requiring sharp dissection | 100 | 0
  requiring extensive sharp dissection | 0 | 0

4. Primary Outcome: Severity of Adhesions at the Left Lateral Site
Description: as for outcome 2
Time Frame: Severity of adhesions data will be collected during approximately the first 30-60 minutes of the second staged surgery
Measure: Number; unit: percentage of participants
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
percentage of participants
  no adhesions | 0 | 8.3
  filmy and avascular | 0 | 50.0
  requiring blunt dissection | 0 | 8.3
  requiring sharp dissection | 87.5 | 33.3
  requiring extensive sharp dissection | 12.5 | 0

5. Primary Outcome: Severity of Adhesions at the Right Lateral Site
Description: as for outcome 2
Time Frame: Severity of adhesions data will be collected during approximately the first 30-60 minutes of the second staged surgery
Measure: Number; unit: percentage of participants
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
percentage of participants
  no adhesions | 0 | 6.3
  filmy and avascular | 0 | 25.0
  requiring blunt dissection | 7.7 | 50.0
  requiring sharp dissection | 53.8 | 18.8
  requiring extensive sharp dissection | 38.5 | 0.0

6. Primary Outcome: Post-operative Bleeding
Description: Post-operative bleeding through surgical site drainage output.
Time Frame: Post-operative bleeding data will be collected on average, during the first 36 hours after the surgery
Population: The difference in the number of participants analyzed and the total number of participants is due to the information not being properly collected at the time of the surgery. Because there was a lack of confidence in the data, it was discarded.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 13 | 14
cm^3 | 106.38 (78.539) | 108.64 (116.449)

7. Primary Outcome: Adhesion Burden
Description: Skin to bypass time as an indicator of adhesion burden.
Time Frame: Time it takes for patient to be put on bypass (an average time between 0 and 120 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 14 | 16
minutes | 37.39 (10.445) | 23.44 (6.366)

8. Secondary Outcome: Hospital Stay
Description: Number of days post surgery.
Time Frame: Length of stay after second surgery up to 1 month
Population: The difference in the number of participants analyzed and the total number of participants is due to feeding issues unrelated to the surgery or the device that required the subject to remain hospitalized longer than anticipated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Number analyzed (Participants) | 12 | 14
days | 4.75 (2.832) | 6.29 (5.269)

ADVERSE EVENTS:
Arm/Group | No CoSeal Surgical Spray | CoSeal Spray Group
Serious Adverse Events (participants affected / at risk) | 1/16 | 3/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No CoSeal Surgical Spray (N=16) | CoSeal Spray Group (N=19)
Cardiac Arrest unrelated to device (Congenital, familial and genetic disorders) | 1 (1) | 3 (3) — Cardiac Arrest related to complex congenital heart disease which has a 10% mortality rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No